CLINICAL TRIAL: NCT01252628
Title: Phase 1/2 Study of PX-866 and Cetuximab
Brief Title: Phase 1 and 2 Study of PX-866 and Cetuximab
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cascadian Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Organization: Seagen Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PX-866-003
Record Dates: First submitted 2010-12-01; First posted 2010-12-03 (Estimated); Last update posted 2018-05-16 (Actual); Status verified 2015-06

CONDITIONS: Incurable Metastatic Colorectal Carcinoma; Incurable Progressive, Recurrent or Metastatic Squamous Cell Carcinoma of the Head and Neck
Keywords: CRC; SCCHN; PX-866; Cetuximab; ERBITUX; Colon; Head and Neck; Colorectal cancer; Squamous cell carcinoma; PI-3K; PI3 kinase; PI3K
MeSH Terms: conditions — Recurrence; Colorectal Neoplasms; Carcinoma, Squamous Cell; Hereditary Sensory and Autonomic Neuropathies | interventions — PX-866; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- PX-866 (SCCHN) (Experimental): Phase 2 (Squamous Cell Carcinoma of the Head and Neck)
  Interventions: Drug: PX-866 (SCCHN); Drug: Cetuximab (SCCHN)
- Cetuximab (SCCHN) (Active Comparator): Phase 2 (Squamous Cell Carcinoma of the Head and Neck)
  Interventions: Drug: Cetuximab (SCCHN)
- PX-866 (CRC) (Experimental): Phase 2 (Colorectal Carcinoma)
  Interventions: Drug: PX-866 (CRC); Drug: Cetuximab (CRC)
- Cetuximab (CRC) (Active Comparator): Phase 2 (Colorectal Carcinoma)
  Interventions: Drug: Cetuximab (CRC)

INTERVENTIONS:
Drug: PX-866 (SCCHN) — PX-866 administered at the MTD/RD in combination in patients administered weekly on a 21 day cycle.
  Arms: PX-866 (SCCHN)
Drug: Cetuximab (SCCHN) — Cetuximab administered weekly on a 21 day cycle, as standard of care in patients.
  Other Names: Erbitux
  Arms: Cetuximab (SCCHN); PX-866 (SCCHN)
Drug: PX-866 (CRC) — PX-866 administered at the MTD/RD in combination in patients administered weekly on a 21 day cycle.
  Arms: PX-866 (CRC)
Drug: Cetuximab (CRC) — Cetuximab administered weekly on a 21 day cycle in patients, as standard of care.
  Other Names: Erbitux
  Arms: Cetuximab (CRC); PX-866 (CRC)

SUMMARY:
The purpose of this Phase 1/2 open-label study is to determine the safety and efficacy of a cetuximab and PX-866 combination treatment. In the Phase 1 part of the study, the dose of PX-866 to be given in combination with cetuximab will be determined in patients with incurable metastatic CRC or incurable progressive, recurrent or metastatic SCCHN. The Phase 2 part of the study is a randomized evaluation of the antitumor activity and safety of PX-866 in combination with cetuximab versus cetuximab alone in patients with either incurable metastatic CRC who have a history of progression or recurrence following prior irinotecan and oxaliplatin containing regimens or are intolerant of irinotecan (Group 1) or incurable progressive, recurrent or metastatic SCCHN (Group 2).

DETAILED DESCRIPTION:
Phase 1 will determine the maximally tolerated or recommended dose of PX-866 to be given orally on Days 1-21 in combination with cetuximab 250 mg/m2 administered IV weekly on Days 1, 8, and 15 of a 21-day cycle. All patients will receive an initial loading dose of 400 mg/m2 cetuximab rather than 250 mg/m2 on Cycle 1 Day 1. Patients may receive premedication with an H1 antagonist per the cetuximab package insert. Up to 3 dose levels of PX-866 will be evaluated to determine the MTD/RD in cohorts of up to 6 patients using a standard 3+3 dose-escalation design. At least 6 patients will be treated at the MTD/RD. All patients in Phase 1 will be required to undergo PK assessments during Cycle 1 Week 3 to measure cetuximab levels. Exploratory PD assessments will include evaluation of changes in levels of fasting C-peptide as well as changes in EGFR and PI-3K signaling pathways in peripheral blood mononuclear cells (PBMC) and platelets. Additional optional evaluations will include changes in EGFR and PI-3K signaling in paired tumor biopsies provided before and after one cycle of treatment. All patients will be asked, but not required, to provide an archived tumor biopsy sample for evaluation for potential biomarkers of response to PX-866 and cetuximab.

Phase 2 is an open-label, randomized evaluation of the antitumor activity and safety of PX-866 administered orally or via PEG tube (if applicable) at the MTD/RD in combination with cetuximab, versus cetuximab alone in cetuximab-naïve patients with incurable metastatic CRC who have a history of progression or recurrence following prior irinotecan and oxaliplatin containing regimens or are intolerant of irinotecan (Group 1) or patients with incurable progressive, recurrent or metastatic SCCHN (Group 2). Seventy two evaluable patients (36 patients per arm) will be evaluated per indication. Patients will be randomized 1:1 to receive PX-866 + cetuximab or cetuximab alone.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years at time of consent
* Use of a medically accepted form of contraception from the time of consent to completion of all follow-up study visits
* If female of child-bearing potential, negative pregnancy test
* Signed an informed consent
* Measurable disease per Response Evaluation Criteria In Solid Tumors (RECIST)
* Documentation available for last prior systemic treatment including dates of treatment, best response to treatment, duration of best response, and reason for discontinuation of treatment
* Eastern Cooperative Oncology Group (ECOG) 0 or 1
* Group 1: Patients with incurable metastatic CRC with a history of progression or recurrence following prior irinotecan and oxaliplatin containing regimens. Patients who have a history of intolerance of irinotecan based therapy or ineligibility to receive irinotecan are also eligible as long as they have received a prior oxaliplatin containing regimen.
* Group 2: Patients with incurable SCCHN with a history of progression or recurrence following at least one prior platinum based chemotherapy or chemotherapy/radiation containing regimen. Patients who have a history of intolerance of platinum based therapy or history of ineligibility to receive a platinum based regimen are also eligible. SCCHN patients who received cetuximab as a radiosensitizer for locally advanced disease and completed treatment at least 6 months prior to start of study drug treatment are eligible
* In the opinion of the clinical investigator, life expectancy of greater than 3 months
* Adequate hematologic function
* Adequate hepatic function
* Creatinine level ≤1.5 x ULN
* Serum magnesium ≥ LLN.

Exclusion Criteria:

* Has medical, social, or psychosocial factors that, in the opinion of the investigator, could impact safety or compliance with study procedures
* Is breastfeeding
* Treatment with any systemic chemotherapy, epidermal growth factor receptor (EGFR) inhibitor, radiation or experimental agent within 4 weeks of study drug dosing
* Received prior cetuximab, except as defined in inclusion criteria
* Previous treatment with a phosphatidylinositol 3-kinase (PI-3K) inhibitor
* Known human immunodeficiency virus (HIV)
* Poorly controlled diabetes mellitus (IFCC-HbA1C ≥ 53 mmol/mol or DCCT -HbA1C ≥ 7%)
* Kras mutation in codon 12 or 13 (CRC patients only)
* Known or suspected clinically active brain metastases. Previously treated and stable brain metastases are allowable. Stable brain metastases are defined as no change on CT scan or MRI for minimum of two months AND no change in steroid dose for a minimum of four weeks, unless change due to intercurrent infection or other acute event)
* Any other significant medical or psychiatric condition that in the opinion of the investigator renders the patient inadequate for participation
* History of severe hypersensitivity to cetuximab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 2010-12; Primary Completion 2013-11 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
The evaluation of antitumor effects of PX-866 in combination with cetuximab versus cetuximab in patients with incurable metastatic colorectal cancer and/or patients with incurable progressive, recurrent or metastatic SCC of the head and neck. | 21 days

CONTACTS AND LOCATIONS:
Overall Officials: Diana Hausman, MD, Study Director — Cascadian Therapeutics Inc.
Locations (40):
- United States (31):
  - Birmingham Hematology and Oncology Assocs., Birmingham, Alabama
  - University of Alabama Birmingham, Birmingham, Alabama
  - Southwest Cancer Care, Escondido, California
  - Monterey Bay Oncology, Monterey, California
  - Ventura County Hematology Oncology Specialists, Oxnard, California
  - University of Colorado Denver, Aurora, Colorado
  - Rocky Mountain Cancer Centers, Denver, Colorado
  - Eastern Colorado Health Care System - (Denver VA), Denver, Colorado
  - George Washington University - Medical Faculty Associates, Washington D.C., District of Columbia
  - Integrated Community Oncology Network, Jacksonville, Florida
  - Advanced Medical Specialties, Miami, Florida
  - Pasco Pinellas Cancer Center, New Port Richey, Florida
  - Peachtree Hematology-Oncology Consultants, Atlanta, Georgia
  - Center for Cancer and Blood Disorders, Bethesda, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - Saint Louis Cancer Care LLP, Bridgeton, Missouri
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Northwest Cancer Specialists, P.C., Tualatin, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - MUSC Hollings Cancer Center, Charleston, South Carolina
  - Mary Crowley Cancer Center, Dallas, Texas
  - Texas Oncology - Baylor Charles A. Sammons, Dallas, Texas
  - Texas Oncology - Fort Worth, Fort Worth, Texas
  - Texas Oncology - Seton Williamson, Round Rock, Texas
  - Virginia Cancer Specialists, PC, Fairfax, Virginia
  - Peninsula Cancer Institute, Newport News, Virginia
  - Virginia Oncology Associates, Newport News, Virginia
  - Oncology and Hematology Associates of Southwest Virginia, Roanoke, Virginia
  - Columbia Basin Hematology and Oncology, Kennewick, Washington
  - Medical Oncology Associates, Spokane, Washington
- Canada (9):
  - Cross Cancer Institute, Edmonton, Alberta
  - British Columbia Cancer Agency - Vancouver Centre, Vancouver, British Columbia
  - Royal Victoria Regional Health Centre, Barrie, Ontario
  - Northeast Cancer Centre of Health Sciences North, Greater Sudbury, Ontario
  - London Regional Cancer Program, London, Ontario
  - Thunder Bay Regional Health Sciences Centre, Thunder Bay, Ontario
  - Hôpital Charles-LeMoyne, Greenfield Park, Quebec
  - Cité de la Santé de Laval, Laval, Quebec
  - Maisonneuve-Rosemont Hospital Research Centre, Montreal, Quebec